CLINICAL TRIAL: NCT00721305
Title: Antiretroviral Effect of Lovastatin on HIV-1-infected Individuals Without Highly Active Antiretroviral Therapy (HAART): A Phase-II Randomized Clinical Trial (RCT)
Brief Title: Lovastatin: Immunomodulatory Value Evaluation
Acronym: LIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government); Laboratorio Clínico Congregación Mariana (Other); Laboratorios Laproff S.A. (Industry); Humax Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Carlos Julio Montoya Guarin, Associated Professor, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COLCIENCIAS 111540820508
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-09

CONDITIONS: HIV Seropositivity
Keywords: Type 1 human immunodeficiency virus infection; Lovastatin; Adaptive Immunity; Cellular cholesterol; Rho GTPases; Lymphocyte function-associated antigen-1
MeSH Terms: conditions — HIV Seropositivity | interventions — Lovastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): In this arm, subjects will receive 40 mg of Lovastatin (2 tablets of 20 mg each, p.o.), in a daily doses, during twelve months
  Interventions: Drug: Lovastatin
- 2 (Placebo Comparator): In this arm, subjects will receive placebo (2 tablets which will look externally identical to lovastatin: wrapped in the same way, with the same size, shape and color)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Lovastatin — Lovastatin 40 mg daily (2 tablets of 20 mg each, p.o.), during twelve months until the end of the study, or before the end of the study if any AIDS defining disease or toxicity appear
  Other Names: statin
  Arms: 1
Other: placebo — Placebo will be administered daily (2 tablets which will look externally identical to intervention: wrapped in the same way, with the same size, shape and color), during twelve months until the end of the study, or before the end of the study if any AIDS defining disease or toxicity appear
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the long-term administration of statins may benefit the clinical and immunological evolution in HIV-1-infected individuals before the use of antiretroviral therapy is required.

DETAILED DESCRIPTION:
Despite the fact that HAART produces a decrease in HIV-1 replication and plasma HIV-1 RNA levels, and allows an increase in the CD4 T-cell count that leads to a diminution in the incidence of opportunistic infections and mortality, the cost and complexity of HAART regimens, the growing list of long-term side effects, and the eventual development of resistance have underscored the immediate need for additional therapeutic approaches. Statins exert pleiotropic effects through a variety of mechanisms, among which there are several immunological effects that are related and unrelated to their cholesterol-lowering activity. HIV-1 requires cholesterol and lipid rafts for several key stages of its replication cycle; statins-mediated depletion of cholesterol alters the capacity of a cell to form lipid rafts and decreases the HIV-1 infectivity. On the other hand, statins may exert significant modulator effects in the balance of the cytokine network, and alter the activity of Rho GTPases and LFA-1 and ICAM-1 adhesion molecules. Preliminary studies showed that statins (Lovastatin) had anti HIV-1 activity, and that its administration was safe and efficient to control HIV-1 infection in chronically infected individuals who did not receive HAART (in terms of decreasing viral load and increasing CD4 T-cell count). Because very limited clinical data are available on this topic, this study will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic HIV-1 seropositive individuals, with age ≥ 18 years, who are HAART naive
* HIV-1 infection confirmed by:

  * positive Western-blot test dated at least six months before admission to the study;
  * a Western-blot test within the last six months, which was also positive for the p31 and p66 bands
* Detectable viral load < 100,000 copies/ml
* CD4+ T cell count ≥ 350 cells/ul

Exclusion Criteria:

* Inability or unwillingness of patients to give written informed consent.
* Main residence outside Medellin and its metropolitan area, or any indication of difficulties in the follow-up period
* Participation in other clinical trials
* Evidence that the patient will exhibit low adherence to intervention and follow-up (Morisky-Green test)
* Pregnancy or breastfeeding
* Any type of antiretroviral treatment before admission to the study, and therapy with lipid-lowering drugs during the last six months
* Antecedents of allergy, contraindications or intolerance to statins
* Patients receiving medications which can generate relevant interactions with lovastatin: clarithromycin, erythromycin, azithromycin, itraconazole, ketoconazole, nefodozone, cimetidine, rifampin, phenobarbital, carbamazepine, phenytoin.
* Unwillingness to avoid the consumption of Citrus paradise (grapefruit juice) or Saint John's Wort (Hypericum)
* Opportunistic infections or any type of AIDS-defining disease
* Chronic active hepatitis (B or C)
* Any hepatocellular disease, indicated by elevation of liver enzymes (AST or ALT) more than twice the reference value
* Renal failure, indicated by serum creatinine ≥ 2 mg/dl
* Myopathy, indicated by an elevation of creatine phosphokinase (CPK) more than five times the reference values
* Infection or acute disease that requires in-patient treatment
* Active substance-related disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2008-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
1. HIV-1 viral load measured as RNA copies per ml of peripheral blood 2. CD4 T-cell count measured as cells per ul of peripheral blood | Before, 6 and twelve months after the intervention

SECONDARY OUTCOMES:
CD8+ T cell count, CD4/CD8 ratio, Expression of CD38 and HLA-DR, Total serum cholesterol, Cellular cholesterol, Activity of LFA-1 and ICAM-1, Activity of Rho GTPases, Monthly frequency of AIDS defining diseases, hospitalization and mortality | Before, 6 and twelve months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Carlos J Montoya, MD, PhD, Principal Investigator — Universidad de Antioquia; Maria T Rugeles, PhD, Study Chair — Universidad de Antioquia; Fabian A Jaimes, MD, PhD, Study Director — Universidad de Antioquia
Locations (1):
- Group of Immunovirology, Research Universitary Center, University of Antioquia, Medellín, Antioquia, Colombia

REFERENCES:
- [Background] UNAIDS and WHO. AIDS epidemic update 2004. Geneva, Switzerland: Joint United Nations Programme on HIV/AIDS (UNAIDS) and World Health Organization (WHO); 2004 December 2004
- [Background] Instituto Nacional de Salud. Programa Nacional de Prevención y control ITS/SIDA. Colombia 1983-2002. Bogotá: Instituto Nacional de Salud, Ministerio de Salud de la República de Colombia; 2003
- [Background] Cohen DE, Walker BD. Human immunodeficiency virus pathogenesis and prospects for immune control in patients with established infection. Clin Infect Dis. 2001 Jun 15;32(12):1756-68. doi: 10.1086/320759. Epub 2001 May 16. PMID 11360218
- [Background] Giorgi JV, Liu Z, Hultin LE, Cumberland WG, Hennessey K, Detels R. Elevated levels of CD38+ CD8+ T cells in HIV infection add to the prognostic value of low CD4+ T cell levels: results of 6 years of follow-up. The Los Angeles Center, Multicenter AIDS Cohort Study. J Acquir Immune Defic Syndr (1988). 1993 Aug;6(8):904-12. PMID 7686224
- [Background] Hazenberg MD, Otto SA, van Benthem BH, Roos MT, Coutinho RA, Lange JM, Hamann D, Prins M, Miedema F. Persistent immune activation in HIV-1 infection is associated with progression to AIDS. AIDS. 2003 Sep 5;17(13):1881-8. doi: 10.1097/00002030-200309050-00006. PMID 12960820
- [Background] Palella FJ Jr, Delaney KM, Moorman AC, Loveless MO, Fuhrer J, Satten GA, Aschman DJ, Holmberg SD. Declining morbidity and mortality among patients with advanced human immunodeficiency virus infection. HIV Outpatient Study Investigators. N Engl J Med. 1998 Mar 26;338(13):853-60. doi: 10.1056/NEJM199803263381301. PMID 9516219
- [Background] Finzi D, Hermankova M, Pierson T, Carruth LM, Buck C, Chaisson RE, Quinn TC, Chadwick K, Margolick J, Brookmeyer R, Gallant J, Markowitz M, Ho DD, Richman DD, Siliciano RF. Identification of a reservoir for HIV-1 in patients on highly active antiretroviral therapy. Science. 1997 Nov 14;278(5341):1295-300. doi: 10.1126/science.278.5341.1295. PMID 9360927
- [Background] Aberg JA, Zackin RA, Brobst SW, Evans SR, Alston BL, Henry WK, Glesby MJ, Torriani FJ, Yang Y, Owens SI, Fichtenbaum CJ; ACTG 5087 Study Team. A randomized trial of the efficacy and safety of fenofibrate versus pravastatin in HIV-infected subjects with lipid abnormalities: AIDS Clinical Trials Group Study 5087. AIDS Res Hum Retroviruses. 2005 Sep;21(9):757-67. doi: 10.1089/aid.2005.21.757. PMID 16218799
- [Background] Calza L, Manfredi R, Chiodo F. Statins and fibrates for the treatment of hyperlipidaemia in HIV-infected patients receiving HAART. AIDS. 2003 Apr 11;17(6):851-9. doi: 10.1097/00002030-200304110-00010. PMID 12660532
- [Background] Fehr T, Kahlert C, Fierz W, Joller-Jemelka HI, Riesen WF, Rickli H, Wuthrich RP, Ammann P. Statin-induced immunomodulatory effects on human T cells in vivo. Atherosclerosis. 2004 Jul;175(1):83-90. doi: 10.1016/j.atherosclerosis.2004.02.016. PMID 15186950
- [Background] Yilmaz A, Reiss C, Tantawi O, Weng A, Stumpf C, Raaz D, Ludwig J, Berger T, Steinkasserer A, Daniel WG, Garlichs CD. HMG-CoA reductase inhibitors suppress maturation of human dendritic cells: new implications for atherosclerosis. Atherosclerosis. 2004 Jan;172(1):85-93. doi: 10.1016/j.atherosclerosis.2003.10.002. PMID 14709361
- [Background] Kwak B, Mulhaupt F, Veillard N, Pelli G, Mach F. The HMG-CoA reductase inhibitor simvastatin inhibits IFN-gamma induced MHC class II expression in human vascular endothelial cells. Swiss Med Wkly. 2001 Jan 27;131(3-4):41-6. doi: 10.4414/smw.2001.06144. PMID 11219190
- [Background] Liao Z, Cimakasky LM, Hampton R, Nguyen DH, Hildreth JE. Lipid rafts and HIV pathogenesis: host membrane cholesterol is required for infection by HIV type 1. AIDS Res Hum Retroviruses. 2001 Jul 20;17(11):1009-19. doi: 10.1089/088922201300343690. PMID 11485618
- [Background] Del Real G, Jimenez-Baranda S, Lacalle RA, Mira E, Lucas P, Gomez-Mouton C, Carrera AC, Martinez-A C, Manes S. Blocking of HIV-1 infection by targeting CD4 to nonraft membrane domains. J Exp Med. 2002 Aug 5;196(3):293-301. doi: 10.1084/jem.20020308. PMID 12163558
- [Background] del Real G, Jimenez-Baranda S, Mira E, Lacalle RA, Lucas P, Gomez-Mouton C, Alegret M, Pena JM, Rodriguez-Zapata M, Alvarez-Mon M, Martinez-A C, Manes S. Statins inhibit HIV-1 infection by down-regulating Rho activity. J Exp Med. 2004 Aug 16;200(4):541-7. doi: 10.1084/jem.20040061. PMID 15314078
- [Background] Giguere JF, Tremblay MJ. Statin compounds reduce human immunodeficiency virus type 1 replication by preventing the interaction between virion-associated host intercellular adhesion molecule 1 and its natural cell surface ligand LFA-1. J Virol. 2004 Nov;78(21):12062-5. doi: 10.1128/JVI.78.21.12062-12065.2004. PMID 15479847
- [Background] Hakamada-Taguchi R, Uehara Y, Kuribayashi K, Numabe A, Saito K, Negoro H, Fujita T, Toyo-oka T, Kato T. Inhibition of hydroxymethylglutaryl-coenzyme a reductase reduces Th1 development and promotes Th2 development. Circ Res. 2003 Nov 14;93(10):948-56. doi: 10.1161/01.RES.0000101298.76864.14. Epub 2003 Oct 16. PMID 14563711
- [Background] Shimada K, Miyauchi K, Daida H. Early intervention with atorvastatin modulates TH1/TH2 imbalance in patients with acute coronary syndrome: from bedside to bench. Circulation. 2004 May 11;109(18):e213-4; author reply e213-4. doi: 10.1161/01.CIR.0000127616.70152.5D. No abstract available. PMID 15136515
- [Background] Youssef S, Stuve O, Patarroyo JC, Ruiz PJ, Radosevich JL, Hur EM, Bravo M, Mitchell DJ, Sobel RA, Steinman L, Zamvil SS. The HMG-CoA reductase inhibitor, atorvastatin, promotes a Th2 bias and reverses paralysis in central nervous system autoimmune disease. Nature. 2002 Nov 7;420(6911):78-84. doi: 10.1038/nature01158. PMID 12422218
- [Background] Illingworth DR, Tobert JA. HMG-CoA reductase inhibitors. Adv Protein Chem. 2001;56:77-114. doi: 10.1016/s0065-3233(01)56003-9. No abstract available. PMID 11329860
- [Background] Garcia PJ. Pleiotropic effects of statins: moving beyond cholesterol control. Curr Atheroscler Rep. 2005 Feb;7(1):34-9. doi: 10.1007/s11883-005-0073-6. PMID 15683600
- [Background] Blanco-Colio LM, Tunon J, Martin-Ventura JL, Egido J. Anti-inflammatory and immunomodulatory effects of statins. Kidney Int. 2003 Jan;63(1):12-23. doi: 10.1046/j.1523-1755.2003.00744.x. PMID 12472764
- [Background] Vanhaecke J, Van Cleemput J, Van Lierde J, Daenen W, De Geest H. Safety and efficacy of low dose simvastatin in cardiac transplant recipients treated with cyclosporine. Transplantation. 1994 Jul 15;58(1):42-5. PMID 8036706
- [Background] Vaughan CJ, Delanty N. Neuroprotective properties of statins in cerebral ischemia and stroke. Stroke. 1999 Sep;30(9):1969-73. doi: 10.1161/01.str.30.9.1969. PMID 10471452
- [Background] Kallen J, Welzenbach K, Ramage P, Geyl D, Kriwacki R, Legge G, Cottens S, Weitz-Schmidt G, Hommel U. Structural basis for LFA-1 inhibition upon lovastatin binding to the CD11a I-domain. J Mol Biol. 1999 Sep 10;292(1):1-9. doi: 10.1006/jmbi.1999.3047. PMID 10493852
- [Background] Issekutz TB. Inhibition of lymphocyte endothelial adhesion and in vivo lymphocyte migration to cutaneous inflammation by TA-3, a new monoclonal antibody to rat LFA-1. J Immunol. 1992 Nov 15;149(10):3394-402. PMID 1358970
- [Background] Wallays G, Ceuppens JL. Ligation of leukocyte function-associated (LFA) molecule-1 provides an accessory signal for T-cell activation with pokeweed mitogen. Scand J Immunol. 1994 Feb;39(2):137-43. doi: 10.1111/j.1365-3083.1994.tb03352.x. PMID 7905204
- [Background] Moncunill G, Negredo E, Bosch L, Vilarrasa J, Witvrouw M, Llano A, Clotet B, Este JA. Evaluation of the anti-HIV activity of statins. AIDS. 2005 Oct 14;19(15):1697-700. doi: 10.1097/01.aids.0000183517.60384.db. PMID 16184043
- [Background] Sklar PA, Masur H, Grubb JR, Voell J, Witek J, Ono A, Freed EO, Maldarelli F. Pravastatin does not have a consistent antiviral effect in chronically HIV-infected individuals on antiretroviral therapy. AIDS. 2005 Jul 1;19(10):1109-11. doi: 10.1097/01.aids.0000174461.31794.50. No abstract available. PMID 15958846
- [Background] Manfredi R, Calza L, Chiodo F. Long-term statin use does not act on the temporal trend of CD4 cell count in patients on virologically effective HAART. AIDS. 2006 Feb 14;20(3):455-7. doi: 10.1097/01.aids.0000199822.49488.50. PMID 16439881
- [Background] Waters L, Stebbing J, Jones R, Mandalia S, Bower M, Stefanovic M, Nelson M, Gazzard B. The effect of statins on HIV rebound and blips. J Acquir Immune Defic Syndr. 2005 Aug 15;39(5):637-8. No abstract available. PMID 16044021
- [Background] Bonnet F, Balestre E, Thiebaut R, Mercie P, Dupon M, Morlat P, Dabis F; Groupe d'Epidemiologie Clinique du SIDA en Aquitaine (GECSA). Fibrates or statins and lipid plasma levels in 245 patients treated with highly active antiretroviral therapy. Aquitaine Cohort, France, 1999-2001. HIV Med. 2004 May;5(3):133-9. doi: 10.1111/j.1468-1293.2004.00200.x. PMID 15139977
- [Background] Benesic A, Zilly M, Kluge F, Weissbrich B, Winzer R, Klinker H, Langmann P. Lipid lowering therapy with fluvastatin and pravastatin in patients with HIV infection and antiretroviral therapy: comparison of efficacy and interaction with indinavir. Infection. 2004 Aug;32(4):229-33. doi: 10.1007/s15010-004-3136-7. PMID 15293079
- [Background] Hulgan T, Sterling TR, Daugherty J, Arbogast PG, Raffanti S, Ray W. Prescribing of contraindicated protease inhibitor and statin combinations among HIV-infected persons. J Acquir Immune Defic Syndr. 2005 Mar 1;38(3):277-82. PMID 15735444
- [Background] Penzak SR, Chuck SK, Stajich GV. Safety and efficacy of HMG-CoA reductase inhibitors for treatment of hyperlipidemia in patients with HIV infection. Pharmacotherapy. 2000 Sep;20(9):1066-71. doi: 10.1592/phco.20.13.1066.35033. PMID 10999499
- [Background] van der Goot FG, Harder T. Raft membrane domains: from a liquid-ordered membrane phase to a site of pathogen attack. Semin Immunol. 2001 Apr;13(2):89-97. doi: 10.1006/smim.2000.0300. PMID 11308292
- [Background] Manes S, del Real G, Lacalle RA, Lucas P, Gomez-Mouton C, Sanchez-Palomino S, Delgado R, Alcami J, Mira E, Martinez-A C. Membrane raft microdomains mediate lateral assemblies required for HIV-1 infection. EMBO Rep. 2000 Aug;1(2):190-6. doi: 10.1093/embo-reports/kvd025. PMID 11265761
- [Background] Moore JP, Trkola A, Dragic T. Co-receptors for HIV-1 entry. Curr Opin Immunol. 1997 Aug;9(4):551-62. doi: 10.1016/s0952-7915(97)80110-0. PMID 9287172
- [Background] Nguyen DH, Taub DD. Inhibition of chemokine receptor function by membrane cholesterol oxidation. Exp Cell Res. 2003 Nov 15;291(1):36-45. doi: 10.1016/s0014-4827(03)00345-8. PMID 14597406
- [Background] Alfsen A, Iniguez P, Bouguyon E, Bomsel M. Secretory IgA specific for a conserved epitope on gp41 envelope glycoprotein inhibits epithelial transcytosis of HIV-1. J Immunol. 2001 May 15;166(10):6257-65. doi: 10.4049/jimmunol.166.10.6257. PMID 11342649
- [Background] Gummuluru S, Rogel M, Stamatatos L, Emerman M. Binding of human immunodeficiency virus type 1 to immature dendritic cells can occur independently of DC-SIGN and mannose binding C-type lectin receptors via a cholesterol-dependent pathway. J Virol. 2003 Dec;77(23):12865-74. doi: 10.1128/jvi.77.23.12865-12874.2003. PMID 14610207
- [Background] Maziere JC, Landureau JC, Giral P, Auclair M, Fall L, Lachgar A, Achour A, Zagury D. Lovastatin inhibits HIV-1 expression in H9 human T lymphocytes cultured in cholesterol-poor medium. Biomed Pharmacother. 1994;48(2):63-7. doi: 10.1016/0753-3322(94)90077-9. PMID 7522603
- [Background] Guyader M, Kiyokawa E, Abrami L, Turelli P, Trono D. Role for human immunodeficiency virus type 1 membrane cholesterol in viral internalization. J Virol. 2002 Oct;76(20):10356-64. doi: 10.1128/jvi.76.20.10356-10364.2002. PMID 12239312
- [Background] Viard M, Parolini I, Sargiacomo M, Fecchi K, Ramoni C, Ablan S, Ruscetti FW, Wang JM, Blumenthal R. Role of cholesterol in human immunodeficiency virus type 1 envelope protein-mediated fusion with host cells. J Virol. 2002 Nov;76(22):11584-95. doi: 10.1128/jvi.76.22.11584-11595.2002. PMID 12388719
- [Background] Vincent N, Genin C, Malvoisin E. Identification of a conserved domain of the HIV-1 transmembrane protein gp41 which interacts with cholesteryl groups. Biochim Biophys Acta. 2002 Dec 23;1567(1-2):157-64. doi: 10.1016/s0005-2736(02)00611-9. PMID 12488049
- [Background] Saez-Cirion A, Nir S, Lorizate M, Agirre A, Cruz A, Perez-Gil J, Nieva JL. Sphingomyelin and cholesterol promote HIV-1 gp41 pretransmembrane sequence surface aggregation and membrane restructuring. J Biol Chem. 2002 Jun 14;277(24):21776-85. doi: 10.1074/jbc.M202255200. Epub 2002 Apr 2. PMID 11929877
- [Background] Campbell SM, Crowe SM, Mak J. Virion-associated cholesterol is critical for the maintenance of HIV-1 structure and infectivity. AIDS. 2002 Nov 22;16(17):2253-61. doi: 10.1097/00002030-200211220-00004. PMID 12441796
- [Background] Liao Z, Graham DR, Hildreth JE. Lipid rafts and HIV pathogenesis: virion-associated cholesterol is required for fusion and infection of susceptible cells. AIDS Res Hum Retroviruses. 2003 Aug;19(8):675-87. doi: 10.1089/088922203322280900. PMID 13678470
- [Background] Lee YM, Liu B, Yu XF. Formation of virus assembly intermediate complexes in the cytoplasm by wild-type and assembly-defective mutant human immunodeficiency virus type 1 and their association with membranes. J Virol. 1999 Jul;73(7):5654-62. doi: 10.1128/JVI.73.7.5654-5662.1999. PMID 10364315
- [Background] Lindwasser OW, Resh MD. Human immunodeficiency virus type 1 Gag contains a dileucine-like motif that regulates association with multivesicular bodies. J Virol. 2004 Jun;78(11):6013-23. doi: 10.1128/JVI.78.11.6013-6023.2004. PMID 15140999
- [Background] Fortin JF, Cantin R, Lamontagne G, Tremblay M. Host-derived ICAM-1 glycoproteins incorporated on human immunodeficiency virus type 1 are biologically active and enhance viral infectivity. J Virol. 1997 May;71(5):3588-96. doi: 10.1128/JVI.71.5.3588-3596.1997. PMID 9094631
- [Background] Nguyen DH, Hildreth JE. Evidence for budding of human immunodeficiency virus type 1 selectively from glycolipid-enriched membrane lipid rafts. J Virol. 2000 Apr;74(7):3264-72. doi: 10.1128/jvi.74.7.3264-3272.2000. PMID 10708443
- [Background] Zheng YH, Plemenitas A, Fielding CJ, Peterlin BM. Nef increases the synthesis of and transports cholesterol to lipid rafts and HIV-1 progeny virions. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8460-5. doi: 10.1073/pnas.1437453100. Epub 2003 Jun 24. PMID 12824470
- [Background] Wang JK, Kiyokawa E, Verdin E, Trono D. The Nef protein of HIV-1 associates with rafts and primes T cells for activation. Proc Natl Acad Sci U S A. 2000 Jan 4;97(1):394-9. doi: 10.1073/pnas.97.1.394. PMID 10618429
- [Background] Albi E, Viola Magni MP. The role of intranuclear lipids. Biol Cell. 2004 Oct;96(8):657-67. doi: 10.1016/j.biolcel.2004.05.004. PMID 15519699
- [Background] Fernandez C, Lobo Md Mdel V, Gomez-Coronado D, Lasuncion MA. Cholesterol is essential for mitosis progression and its deficiency induces polyploid cell formation. Exp Cell Res. 2004 Oct 15;300(1):109-20. doi: 10.1016/j.yexcr.2004.06.029. PMID 15383319
- [Background] Butini L, De Fougerolles AR, Vaccarezza M, Graziosi C, Cohen DI, Montroni M, Springer TA, Pantaleo G, Fauci AS. Intercellular adhesion molecules (ICAM)-1 ICAM-2 and ICAM-3 function as counter-receptors for lymphocyte function-associated molecule 1 in human immunodeficiency virus-mediated syncytia formation. Eur J Immunol. 1994 Sep;24(9):2191-5. doi: 10.1002/eji.1830240939. PMID 7916296
- [Background] Tremblay MJ, Fortin JF, Cantin R. The acquisition of host-encoded proteins by nascent HIV-1. Immunol Today. 1998 Aug;19(8):346-51. doi: 10.1016/s0167-5699(98)01286-9. No abstract available. PMID 9709501
- [Background] Park SW, Royal W 3rd, Semba RD, Wiegand GW, Griffin DE. Expression of adhesion molecules and CD28 on T lymphocytes during human immunodeficiency virus infection. Clin Diagn Lab Immunol. 1998 Jul;5(4):583-7. doi: 10.1128/CDLI.5.4.583-587.1998. PMID 9665971
- [Background] Pearce-Pratt R, Phillips DM. Studies of adhesion of lymphocytic cells: implications for sexual transmission of human immunodeficiency virus. Biol Reprod. 1993 Mar;48(3):431-45. doi: 10.1095/biolreprod48.3.431. PMID 8452921
- [Background] Schrier RD, McCutchan JA, Wiley CA. Mechanisms of immune activation of human immunodeficiency virus in monocytes/macrophages. J Virol. 1993 Oct;67(10):5713-20. doi: 10.1128/JVI.67.10.5713-5720.1993. PMID 8371336
- [Background] Fujiwara M, Tsunoda R, Shigeta S, Yokota T, Baba M. Human follicular dendritic cells remain uninfected and capture human immunodeficiency virus type 1 through CD54-CD11a interaction. J Virol. 1999 May;73(5):3603-7. doi: 10.1128/JVI.73.5.3603-3607.1999. PMID 10196251
- [Background] Tsunetsugu-Yokota Y, Yasuda S, Sugimoto A, Yagi T, Azuma M, Yagita H, Akagawa K, Takemori T. Efficient virus transmission from dendritic cells to CD4+ T cells in response to antigen depends on close contact through adhesion molecules. Virology. 1997 Dec 22;239(2):259-68. doi: 10.1006/viro.1997.8895. PMID 9434717
- [Background] Hioe CE, Chien PC Jr, Lu C, Springer TA, Wang XH, Bandres J, Tuen M. LFA-1 expression on target cells promotes human immunodeficiency virus type 1 infection and transmission. J Virol. 2001 Jan;75(2):1077-82. doi: 10.1128/JVI.75.2.1077-1082.2001. PMID 11134324
- [Background] Hildreth JE, Orentas RJ. Involvement of a leukocyte adhesion receptor (LFA-1) in HIV-induced syncytium formation. Science. 1989 Jun 2;244(4908):1075-8. doi: 10.1126/science.2543075.
- [Background] Graaf MR, Richel DJ, van Noorden CJ, Guchelaar HJ. Effects of statins and farnesyltransferase inhibitors on the development and progression of cancer. Cancer Treat Rev. 2004 Nov;30(7):609-41. doi: 10.1016/j.ctrv.2004.06.010. PMID 15531395
- [Background] Raggatt LJ, Partridge NC. HMG-CoA reductase inhibitors as immunomodulators: potential use in transplant rejection. Drugs. 2002;62(15):2185-91. doi: 10.2165/00003495-200262150-00002. PMID 12381218
- [Background] Leung BP, Sattar N, Crilly A, Prach M, McCarey DW, Payne H, Madhok R, Campbell C, Gracie JA, Liew FY, McInnes IB. A novel anti-inflammatory role for simvastatin in inflammatory arthritis. J Immunol. 2003 Feb 1;170(3):1524-30. doi: 10.4049/jimmunol.170.3.1524. PMID 12538717
- [Background] McKay A, Leung BP, McInnes IB, Thomson NC, Liew FY. A novel anti-inflammatory role of simvastatin in a murine model of allergic asthma. J Immunol. 2004 Mar 1;172(5):2903-8. doi: 10.4049/jimmunol.172.5.2903. PMID 14978092
- [Background] Pasternak RC, Smith SC Jr, Bairey-Merz CN, Grundy SM, Cleeman JI, Lenfant C; American College of Cardiology; American Heart Association; National Heart, Lung and Blood Institute. ACC/AHA/NHLBI clinical advisory on the use and safety of statins. J Am Coll Cardiol. 2002 Aug 7;40(3):567-72. doi: 10.1016/s0735-1097(02)02030-2. No abstract available. PMID 12142128
- [Background] Liao Z, Roos JW, Hildreth JE. Increased infectivity of HIV type 1 particles bound to cell surface and solid-phase ICAM-1 and VCAM-1 through acquired adhesion molecules LFA-1 and VLA-4. AIDS Res Hum Retroviruses. 2000 Mar 1;16(4):355-66. doi: 10.1089/088922200309232. PMID 10716373
- [Background] Liang KY, Zeger SL. Regression analysis for correlated data. Annu Rev Public Health. 1993;14:43-68. doi: 10.1146/annurev.pu.14.050193.000355. No abstract available. PMID 8323597
- [Derived] Montoya CJ, Higuita EA, Estrada S, Gutierrez FJ, Amariles P, Giraldo NA, Jimenez MM, Velasquez CP, Leon AL, Rugeles MT, Jaimes FA. Randomized clinical trial of lovastatin in HIV-infected, HAART naive patients (NCT00721305). J Infect. 2012 Dec;65(6):549-58. doi: 10.1016/j.jinf.2012.10.016. Epub 2012 Oct 17. PMID 23085245
- [Derived] Montoya CJ, Jaimes F, Higuita EA, Convers-Paez S, Estrada S, Gutierrez F, Amariles P, Giraldo N, Penaloza C, Rugeles MT. Antiretroviral effect of lovastatin on HIV-1-infected individuals without highly active antiretroviral therapy (The LIVE study): a phase-II randomized clinical trial. Trials. 2009 Jun 18;10:41. doi: 10.1186/1745-6215-10-41. PMID 19538732